CLINICAL TRIAL: NCT02098941
Title: A Retrospective Study to Evaluate Retention Rate of Topiramate With That of Levetiracetam and Oxcarbazepine in a Long-term Epilepsy Treatment
Brief Title: Evaluate Retention Rate of Topiramate, Levetiracetam and Oxcarbazepine in a Long-term Epilepsy Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Principal Investigator, Sang Kun Lee, Professor, Seoul National University Hospital
Other Study IDs: 0620133760
Record Dates: First submitted 2014-03-19; First posted 2014-03-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Epilepsy
Keywords: topiramate; oxcarbazepine; levetiracetam; retention rate
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Topiramate: Subjects who newly visited to the investigator institution during January 1st 2006 to December 31st of 2010 and began their treatment with topiramate as mono or add-on therapy with conventional drugs.
- Levetiracetam: Subjects who newly visited to the investigator institution during January 1st 2006 to December 31st of 2010 and began their treatment with levetiracetam as mono or add-on therapy with conventional drugs.
- Oxcarbazepine: Subjects who newly visited to the investigator institution during January 1st 2006 to December 31st of 2010 and began their treatment with oxcarbazepine as mono or add-on therapy with conventional drugs.

SUMMARY:
The Objective of this study is to compare 2-year retention rate of topiramate, levetiracetam and oxcarbazepine in a long term epilepsy treatment.

DETAILED DESCRIPTION:
Primary objective The Objective of this study is to compare 2-year retention rate of topiramate, levetiracetam and oxcarbazepine in a long term epilepsy treatment.

Secondary objective The main secondary objective of this study is to evaluate confounding factors associated with retention rate of topiramate compared with other anticonvulsants.

1. Baseline characteristics

   * Seizure Type
   * Gender
   * Age of onset
2. Treatment regimen

   * Number of concomitant medication
   * Type of drug combination
   * Final target dose
   * Titration speed

Other secondary objectives

The other secondary objectives of this study are to compare followings by each medication:

* Rate of seizure reduction (≥75%, ≥50%)
* Rate of seizure freedom

ELIGIBILITY:
Inclusion Criteria:

* Subjects who began their treatment with topiramate, levetiracetam or oxcarbazepine as mono or add-on therapy with conventional drugs.
* Subjects who are with partial or generalized epilepsy

Exclusion Criteria:

* Subjects who administered combination therapy in topiramate, levetiracetam or oxcarbazepine
* Subjects who have past experience of surgery for epilepsy treatment
* Subjects who were not followed up for at least 1 year

Ages: 15 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who newly visited to epilepsy center in a tertiary hospital during January 1st 2006 to December 31st of 2010
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Retention rate of topiramate, levetiracetam and oxcarbazepine during 24 months of treatment | 24months
  Overall retention rates of three treatment groups at two years will be presented in patient number (% of continuation or discontinuation).

SECONDARY OUTCOMES:
Evaluate the confounding factors affecting the retention rate | 24 months
  -Confounding factors associated with retention rate
  : Seizure Type, gender, age, treatment regimen, number of concomitant medication, type of drug combination, final target dose, titration speed
Evaluate the response rate through seizure reduction (≥75%, ≥50%) in 2-year treatment with each antiepileptic drugs (topiramate, levetiracetam, oxcarbazepine) | 24 months

OTHER OUTCOMES:
main reasons of drug discontinuation | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sang Kun Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Ramsay E, Faught E, Krumholz A, Naritoku D, Privitera M, Schwarzman L, Mao L, Wiegand F, Hulihan J; CAPSS-272 Study Group. Efficacy, tolerability, and safety of rapid initiation of topiramate versus phenytoin in patients with new-onset epilepsy: a randomized double-blind clinical trial. Epilepsia. 2010 Oct;51(10):1970-7. doi: 10.1111/j.1528-1167.2010.02670.x. PMID 20633037
- [Background] Peltola J, Peltola M, Auvinen A, Raitanen J, Fallah M, Keranen T. Retention rates of new antiepileptic drugs in localization-related epilepsy: a single-center study. Acta Neurol Scand. 2009 Jan;119(1):55-60. doi: 10.1111/j.1600-0404.2008.01062.x. Epub 2008 Jun 24. PMID 18616622